CLINICAL TRIAL: NCT03094520
Title: Effects of Transcranial Direct Current Stimulation (tDCS) on Gestural-verbal Brain Associations: the Role of Cognitive Embodiment
Brief Title: Cognitive Embodiment Activation by tDCS
Acronym: GEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Agnes Flöel, Prof.Dr.med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: GEST
Record Dates: First submitted 2017-02-24; First posted 2017-03-29 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Healthy Young Adults
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anodal tDCS + semantic, motor, attentional tasks (Experimental): Combination of gestural (subjects have to indicate if the gesture is related to the word), attentional and motor tasks with anodal stimulation
  Interventions: Device: tDCS
- Sham tDCS + semantic, motor, attentional tasks (Sham Comparator): Combination of gestural (subjects have to indicate if the gesture is related to the word), attentional and motor tasks with sham stimulation
  Interventions: Device: sham-tDCS

INTERVENTIONS:
Device: tDCS — Transcranial direct current stimulation (tDCS)
  Other Names: Neuroconn
  Arms: Anodal tDCS + semantic, motor, attentional tasks
Device: sham-tDCS — sham stimulation
  Other Names: Neuroconn
  Arms: Sham tDCS + semantic, motor, attentional tasks

SUMMARY:
The main objective of the proposed research is to extend our understanding of how gesture and language interact, focusing on the role of cognitive embodiment in this interaction, and to explore the neural systems that support links between language and actions systems.

ELIGIBILITY:
Inclusion Criteria:

* Right handedness
* unobtrusive neuropsychological screening

Exclusion Criteria:

* History of severe alcoholism or use of drugs.
* Severe psychiatric disorders such as depression, psychosis (if not in remission) and severe untreated medical problems.
* Contraindication for MRT (claustrophobia, metallic implants, ferromagnetic metals in the body, disorders of thermoregulation, pregnant women).

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
response time in semantic decision task | assessed during stimulation or sham stimulation of semantic decision task (last approximately 10 min) at specific timepoint within 2 weeks
  Comparing response time in semantic decision task under anodal tDCS compared to sham stimulation (change from sham stimulation)
performance in attentional load task | assessed during stimulation or sham stimulation of attentional load task (last approximately 6 min) at specific timepoint within 2 weeks
  Attentional load task: Participants are presented with a 6 positions ring that includes different shapes, they have to press V when they see a square and N when they see a diamond. They will have to ignore any shapes other than square and diamond within the ring or distractors that appear outside the ring.
  Comparing performance in attentional load task under anodal tDCS compared to sham stimulation (change from sham stimulation)
performance in motor task | assessed during stimulation or sham stimulation of motor task (last approximately 4 min) at specific timepoint within 2 weeks
  Motor Task: Participants are presented with a red Box and they have to click a button each time they see it as fast as they can.
  Comparing performance in motor task under anodal tDCS compared to sham stimulation (change from sham stimulation)

SECONDARY OUTCOMES:
Functional connectivity predictors | assessed during baseline testing
  Connectivity as measured by resting-state fMRI during baseline as predictors for performance and tDCS responsiveness
Other cognitive outcomes: change in working memory performance | change in working memory performance from baseline after 30 min (approximately)
  Digit span backward performance assessed before (baseline) and after stimulation to test for tDCS effects on working memory
Other cognitive outcomes: change in Attention performance | change in attention performance from baseline after 30 min (approximately)
  Digit span forward performance assessed before baseline) and after stimulation to test for tDCS effects on attention

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Floeel, Prof, Principal Investigator — Charite Universitätsmedizin
Locations (1):
- Charité, Berlin, Germany

REFERENCES:
- [Background] Cohen-Maximov T, Avirame K, Floel A, Lavidor M. Modulation of Gestural-verbal Semantic Integration by tDCS. Brain Stimul. 2015 May-Jun;8(3):493-8. doi: 10.1016/j.brs.2014.12.001. Epub 2014 Dec 11. PMID 25558040
- [Background] Floel A, Ellger T, Breitenstein C, Knecht S. Language perception activates the hand motor cortex: implications for motor theories of speech perception. Eur J Neurosci. 2003 Aug;18(3):704-8. doi: 10.1046/j.1460-9568.2003.02774.x. PMID 12911767
- [Background] Floel A, Rosser N, Michka O, Knecht S, Breitenstein C. Noninvasive brain stimulation improves language learning. J Cogn Neurosci. 2008 Aug;20(8):1415-22. doi: 10.1162/jocn.2008.20098. PMID 18303984